CLINICAL TRIAL: NCT01675778
Title: Influence of Body Size and Composition on Response to Hydromorphone in ED Patients With Acute Pain
Brief Title: Association Between Body Size and Response to Hydromorphone in ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-445; NCT03789500 (obsolete NCT alias)
Record Dates: First submitted 2012-08-23; First posted 2012-08-30 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: hydromorphone; acute pain; emergency department
MeSH Terms: conditions — Pain; Acute Pain; Emergencies | interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hydromorphone (Other): Every enrolled patients will receive a fixed dose (1mg) of intravenous hydromorphone. Pain scale change, patients' satisfaction, requirements for additional pain medications, side effects and adverse events will be recorded at 15 and 30 minutes. Patients' weight and height will be measured. Age, gender, and race/ethnicity will also be recorded. Blood draw for genetic study will be performed.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: Hydromorphone — a fixed dose (1 mg) of hydromorphone will be given to the study subjects
  Other Names: dilaudid

SUMMARY:
Pain is the most common complaint for patients presenting to the emergency department (ED). Inadequate pain relief is also a common problem in ED. Patients' pain perceptions and responses to intravenous opioids vary widely and are influenced by multiple factors. The objective of the current study is to examine the association between total body weight, BMI (body mass index) and clinical response to a fixed dose of intravenous hydromorphone.

DETAILED DESCRIPTION:
Pain is the most common complaint for patients presenting to the emergency department (ED). Morphine and hydromorphone are the two most commonly administrated intravenous opioid analgesics. However, a large inter-individual variation in the response to morphine or hydromorphone has been observed and a significant number of patients do not have satisfactory pain relief after receiving commonly administered doses of these two medications. Current studies have focused on investigating optimal strategies of intravenous opioid use for moderate and severe pain in the ED.

Contrary to the commonly recommended total body weight (TBW) based dosing strategy, a recent publication did not demonstrate a linear relationship between TBW and clinical response to morphine.

The ultimate goal of the research is to identify optimal methods of dosing opioids to alleviate pain in ED patients. The objective of this study is to examine the association between two measures of body size/body composition and response to a standard dose of hydromorphone. The null hypothesis is that there is no association between the measures of body size/composition and response to 1 mg hydromorphone, and thus no difference between the associations. If a strong association exists between TBW or BMI and pain response, it will lend support for the importance of taking body size or composition into account when making decisions about hydromorphone dosing in the ED. It will lay the groundwork for future studies of analgesic dosing. This is of particular importance given the increasing prevalence of obesity in the US and other developed nations.

Specific Aims:

1. To test the association between analgesic response to a standard dose of hydromorphone and total body weight in ED patients with acute pain requiring intravenous opioid analgesia.
2. To test the association between analgesic response to a standard dose of hydromorphone and BMI.
3. To compare the associations between analgesic response to a standard dose of hydromorphone and the two measures of body size/composition, BMI and TBW.
4. To assess whether the associations between response to hydromorphone and these measures of body size/composition are confounded or modified by gender, age, ethnicity and certain genetic polymorphisms.

The results of the current study will suggest whether body size or composition play a role in the clinical response to hydromorphone and may lay the groundwork for further studies to determine whether dosing should be modified to take these characteristics into account either continuously, e.g. 0.015 mg/kg hydromorphone or categorically (increasing doses by category of BMI).

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Age 18 - 65 years old
* Acute pain (less than 7 days in duration)
* Pain with sufficient severity to warrant use of intravenous opioids in the judgment of ED attending physician

Exclusion Criteria:

* Allergy to hydromorphone
* Systolic blood pressure < 90 mm Hg
* Room air oxygen saturation by pulse oximetry < 95% at baseline without supplemental oxygen
* Alcohol or other drug intoxication as judged by the attending physician
* Suspicion of drug seeking by ED physician
* Use of opioids within the past 24 hours
* Use of a monoamine oxidase inhibitor
* Concurrent use of benzodiazepines
* Presence of a chronic pain syndrome (such as sickle cell disease, peripheral neuropathy, diabetic neuropathy, or fibromyalgia)
* History of COPD, sleep apnea, renal failure, liver disease
* Pregnancy or breast feeding
* Prior entry of patient in the study
* Inability or unwillingness to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Birnbaum, MD, Principal Investigator — Jacobi Medical Center, Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Jacobi Medical Center, The Bronx, New York
  - North Central Bronx Hospital, The Bronx, New York

REFERENCES:
- [Derived] Xia S, Chew E, Choe D, Hernandez L, Birnbaum A. No correlation between body size and hydromorphone analgesia in obese patients in ED. Am J Emerg Med. 2015 Oct;33(10):1522-3. doi: 10.1016/j.ajem.2015.07.020. Epub 2015 Jul 21. No abstract available. PMID 26286816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were patients with acute pain recruited from the Emergency Department at Jacobi Medical Center
Groups:
- Hydromorphone: Every enrolled patients will receive a fixed dose (1mg) of intravenous hydromorphone.
Period: Overall Study
Arm/Group | Hydromorphone
Started | 174
Completed | 174
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 174 participants completed the treatment but only 163 participants were included in data analysis. The 11 participants were excluded from the data analysis because 2 had prior opioid use, 2 had chronic pain instead acute pain and 7 did not get measured or weighed by staff as required.
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Age, Categorical [Count of Participants; unit: Participants] — age
  Participants
    <=18 years | 0
    Between 18 and 65 years | 163
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: year] — age
  year | 39 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — gender
  Participants
    Female | 101
    Male | 62
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 93
  White | 15
  Black or African American | 40
  Asian/Pacific Islander | 8
  Others | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 163
Cause of pain [Count of Participants; unit: Participants]
  Injury | 15
  Noninjury | 148
Pain duration [Median (Inter-Quartile Range); unit: days] | 1 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Change in Pain Intensity and TBW at 30 Minutes Post-treatment
Description: Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported 30 minutes after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and total body weight (TBW). The reported value represents the correlation coefficient.
Time Frame: 30 minutes post-treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient | -0.03 [-0.18 to 0.13]

2. Secondary Outcome: Correlation Between Change in Pain Intensity and TBW at 15 Minutes Post-treatment
Description: Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported 15 minutes after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and total body weight (TBW). The reported value represents the correlation coefficient.
Time Frame: 15 minutes post-treatment
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient | -0.06 [-0.21 to 0.10]

3. Secondary Outcome: Pain Treatment Satisfaction Levels as Assessed by Self-report
Description: Participant's satisfaction with their treatment were assessed by self-report. After treatment, participants were asked "How satisfied are you with the result of your pain treatment today?" and they were told to pick their satisfaction level from "very dissatisfied," "dissatisfied," "uncertain," "satisfied," and "very satisfied." Participants at each level is reported.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants
  Very dissatisfied | 2
  Dissatisfied | 8
  Uncertain | 26
  Satisfied | 68
  Very satisfied | 57
  Missing | 2

4. Secondary Outcome: Number of Participants With Oxygen Saturation Level < 92%
Description: Opioids can induce respiratory depression, which could lead to low oxygen saturation level. Prolonged low oxygen saturation level < 92% could cause brain damage. Understanding all potential negative impacts of Hydromorphone helps make it safer for clinical use.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 1

5. Secondary Outcome: Number of Participants With Nausea
Description: Opioids can could induce nausea. Number of participants with nausea is reported. Understanding all potential negative impacts of Hydromorphone helps make it safer for clinical use.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 33

6. Secondary Outcome: Effect of Gender on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of gender on the correlation between Total Body Weight (TBW) and change in pain intensity. Participants were asked to rate their pain levels from o (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and total body weight (TBW). The reported value represents the correlation coefficient.
Time Frame: 30 minutes post-treatment
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient
  Female | 0.06 [-0.25 to 0.14]
  Male | 0.11 [-0.15 to 0.35]

7. Secondary Outcome: Effects of Race/Ethnicity on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of race/ethnicity on the correlation between total body weight (TBW) and change in pain intensity. Participants were asked to rate their pain levels from o (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and total body weight (TBW). The reported value represents the correlation coefficient.
Time Frame: 30 minutes post-treatment
Population: Only Hispanic and African American were analyzed, since these two populations were most common in our study participants (Hispanic 57.1%; African American 24.5%).
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 133
correlation coefficient
  Hispanic | -0.03 [-0.17 to 0.24]
  African American | 0.08 [-0.24 to 0.38]

8. Secondary Outcome: Effects of Single-nucleotide Polymorphisms of Opioid Receptor (OPRM1, A118G) on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of genetic factors on the correlation between Total Body Weight (TBW) and change in pain intensity. Clinical responses to hydromorphone could be affected by the single-nucleotide polymorphisms (SNPs) in gene involving opioid receptor (OPRM1, A118G). Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. The median and inter-quantile ranges of pain intensity reduction post-treatment were compared among patients by Kruskal-Wallis test.
Time Frame: 30 minutes post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
score on a scale
  AA | 5.0 [3 to 8]
  AG | 7.0 [4 to 8]
  GG | 6.0 [4 to 8.0]

9. Secondary Outcome: Effects of Age on the Correlation Between TBW and Change in Pain Intensity
Description: Age might affect the responses to the hydromorphone treatment. The effects of age on the correlation between total body weight (TBW) and change in pain intensity. The mean of age was compared in TBW tertile groups.
Time Frame: 30 minutes post-treatment
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
years
  low TBW tertile | 39.5 (11.0)
  medium TBW tertile | 42.1 (11.0)
  high TBW tertile | 39.3 (14.1)

10. Other Pre Specified Outcome: Number of Participants Who Desired for More Analgesics
Description: Some participants liked to receive additional analgesics after hydromorphone treatment. Number of participants who desired for additional analgesics is reported.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 37

11. Primary Outcome: Correlation Between Change in Pain Intensity and BMI at 30 Minutes Post-treatment
Description: Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported 30 minutes after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and body mass index (BMI). The reported value represents the correlation coefficient.
Time Frame: 30 minutes post-treatment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient | -0.04 [-0.16 to 0.08]

12. Secondary Outcome: Number of Participant With Systolic Blood Pressure < 90 mmHg
Description: Opioids can induce low blood pressure. Prolonged low systolic blood pressure < 90 mmHg can cause shock and multi-organ failure. Understanding all potential negative impacts of Hydromorphone helps make it safer for clinical use.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 0

13. Secondary Outcome: Effect of Gender on the Correlation Between BMI and Change in Pain Intensity
Description: This study evaluated the effect of gender on the correlation between body mass index (BMI) and change in pain intensity. Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and body mass index (BMI). The reported value represents the correlation coefficient.
Time Frame: 30 minutes post-treatment
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient
  Female | 0.0017 [-0.193 to 0.197]
  Male | 0.1887 [-0.064 to 0.418]

14. Secondary Outcome: Number of Participants With Vomit
Description: Opioids can induce vomit. Number of participants with vomit is reported. Understanding all potential negative impacts of Hydromorphone helps make it safer for clinical use.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 4

15. Secondary Outcome: Number of Participants With Skin Itching
Description: Opioids can induce skin itching. Number of participants with skin itching is reported. Understanding all potential negative impacts of Hydromorphone helps make it safer for clinical use.
Time Frame: 30 minutes post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
Participants | 15

16. Secondary Outcome: Association Between Change in Pain Intensity and BMI at 15 Minutes Post-treatment
Description: Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported 15 minutes after treatment. Pearson correlation was used to assess the correlation between change in pain intensity and body mass index (BMI). The reported value represents the correlation coefficient.
Time Frame: 15 minutes post-treatment
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
correlation coefficient | -0.05 [-0.21 to 0.10]

17. Secondary Outcome: Effects of Single-nucleotide Polymorphisms of Opioid Transporter (ABCB1, C3435T) on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of genetic factors on the correlation between Total Body Weight (TBW) and change in pain intensity. Clinical responses to hydromorphone could be affected by the single-nucleotide polymorphisms (SNPs) in gene involving opioid transporter (ABCB1, C3435T). Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. The mean and inter-quantile ranges of pain intensity reduction post-treatment were compared among patients by Kruskal-Wallis test.
Time Frame: 30 minutes post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
score on a scale
  CC | 5.0 [2 to 7]
  CT | 5.0 [3 to 8]
  TT | 6.0 [3 to 8]

18. Secondary Outcome: Effects of Single-nucleotide Polymorphisms of Pain Sensitivity (COMT, G1947A) on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of genetic factors on the correlation between Total Body Weight (TBW) and change in pain intensity. Clinical responses to hydromorphone could be affected by the single-nucleotide polymorphisms (SNPs) in gene involving pain sensitivity (COMT, G1947A). Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. The mean and inter-quantile ranges of pain intensity reduction post-treatment were compared among patients by Kruskal-Wallis test.
Time Frame: 30 minutes post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
score on a scale
  AA | 5.0 [2 to 8]
  AG | 6.0 [3 to 8]
  GG | 5.0 [3 to 8]

19. Secondary Outcome: Effects of Single-nucleotide Polymorphisms of Opioid Metabolism (UGT2B7, -G840A) on the Correlation Between TBW and Change in Pain Intensity
Description: This study evaluated the effect of genetic factors on the correlation between Total Body Weight (TBW) and change in pain intensity. Clinical responses to hydromorphone could be affected by the single-nucleotide polymorphisms (SNPs) in gene involving opioid metabolism (UGT2B7, -G840A). Participants were asked to rate their pain levels from 0 (=no pain) to 10 (= worst pain). The change in pain intensity was determined by subtracting the intensity reported before treatment from the intensity reported after treatment. The mean and inter-quantile ranges of pain intensity reduction post-treatment were compared among patients by Kruskal-Wallis test.
Time Frame: 30 minutes post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hydromorphone
Number analyzed (Participants) | 163
score on a scale
  AA | 5.0 [3 to 8]
  AG | 5.0 [3 to 8]
  GG | 6.0 [3 to 8]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded till 30 minutes after hydromorphone administration while participants were at the ED.
Description: Oxygen saturation was measured by pule oximetry. Blood pressure was measured by blood pressure monitor. Nausea, vomit, and itching were recorded by direct observation.
Arm/Group | Hydromorphone
All-Cause Mortality (participants affected / at risk) | 0/174
Serious Adverse Events (participants affected / at risk) | 1/174
Other Adverse Events (participants affected / at risk) | 52/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone (N=174)
Oxygen saturation level < 92% (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hydromorphone could cause respiratory depression, which could lead to low oxygen saturation level.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone (N=174)
Nausea (Gastrointestinal disorders) | 33 (33) — Hydromorphone could cause nausea.
Vomit (Gastrointestinal disorders) | 4 (4) — Hydromorphone could cause vomit.
Itching (Skin and subcutaneous tissue disorders) | 15 (15) — Hydromorphone could cause skin itching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes